CLINICAL TRIAL: NCT01334281
Title: A Phase 1, Investigatory Initiated, In-vitro Standardization of B Cell Elispot Assays
Brief Title: An In-vitro Standardization of B Cell Elispot Assays
Status: Terminated | Type: Observational
Why Stopped: Technical difficulties perfecting laboratory test used on blood samples.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Anat Tambur, Director, Transplant Immunology Laboratory, Comprehensive Transplant Center; Research Professor, Feinberg School of Medicine, Northwestern University
Other Study IDs: STU00027653 1682-05; 0037-370-285V-AT (Other: Northwestern University Internal Tracking Number)
Record Dates: First submitted 2009-04-13; First posted 2011-04-13 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Transplant Sensitization; Panel Reactive Antibody; Sensitization to HLA Antigens
Keywords: Panel Reactive Antibody (PRA); Sensitization; Organ Transplant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subjects will serve as a source of B-lineage cells, which will be tested for their ability to produce IgG, tetanus antibodies, (as controls) and HLA specific antibodies that coorespond to those detected by the flow PRA assay. They will be retained until they are used up.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blood: Undergoing Desensitization: Transplant subjects give blood at specified time points. Sensitization to HLA antigens is a barrier to transplant. Several U.S. institutions have protocols for desensitization where patients are treated with IV immunoglobulins (IVIg) and plasmapheresis (PP) to reduce circulating HLA-directed antibody levels. Labs provide doctors information on circulating donor-specific antibody (DSA) levels. These results are the main indicator whether to proceed with transplant. However, no information is given on the fate of the B cells that produce the DSA.
  Interventions: Procedure: Blood Draw
- Blood: NOT Undergoing Desensitization: Transplant subjects give blood at specified time points. Sensitization to HLA antigens is a barrier to transplant. Several U.S. institutions have protocols for desensitization where patients are treated with IV immunoglobulins (IVIg) and plasmapheresis (PP) to reduce circulating HLA-directed antibody levels. Labs provide doctors information on circulating donor-specific antibody (DSA) levels. These results are the main indicator whether to proceed with transplant. However, no information is given on the fate of the B cells that produce the DSA.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Three tubes of blood will be drawn (three 10ml-green top), 7 times (total of 210 ml for study) at the indicated time points: 1) enrollment, 2) anticipated midpoint of desensitization, 3) prior to transplant, 4) three months post-transplant, 5) six months post-transplant, 6) 12 months post-transplant, and 7) 24 months post-transplant.
  Groups: Blood: Undergoing Desensitization
Procedure: Blood Draw — Three tubes of blood will be drawn (three 10ml-green top) twice (60 ml total for study), 8-12 weeks apart. Can be drawn during clinic visit or separate standard of care dialysis visit.
  Groups: Blood: NOT Undergoing Desensitization

SUMMARY:
This study is being done because the study doctor is trying to develop a new test which will help transplant doctors monitor patients with high panel reactive antibodies (PRA). The test would be used to monitor patients' PRA when doctors are trying to lower it through a process known as desensitization. Desensitization lowers high PRA levels and allows patients to receive transplants. This is a single center study to evaluate and optimize the use of a new laboratory test to detect and measure the immune system's functioning.

DETAILED DESCRIPTION:
Sensitization to HLA antigens is the main barrier to solid organ transplantation. Currently, HLA sensitization is monitored by testing patients' serum against a panel of HLA antigens (whether those will be presented on cell surface or on solid phase matrixes) and calculating the % of positive responses. Such result give indication of the relative breadth of sensitization but not on it "depth" - the relative strength of specific antibodies, nor does it provide any information regarding the memory B cells / plasma cells that can manufacture a specific HLA directed antibody.

This is a single center study to evaluate and optimize the use of in-vitro assay to enumerate B cells producing human leukocyte antigens (HLA)-specific antibodies. The proposed assay is based on principles used for enumeration of specific cytokine producing memory T cells - an ELISPOT assay. The investigators are currently using the T cell ELISPOT assay in our laboratory.

The investigators believe that the proposed assay will provide biologically relevant immune measures that are crucial for the long term outcome of transplantation in highly sensitized patients.

Highly sensitized patients encompass a high risk patient group among transplant recipients. The proposed assay is designed to predict the fate of DSA producing (or capable of producing) memory and plasma cells. Thus, it should allow prediction and early detection of activation of the humoral arm of the immune system, specifically against the donor. This, in turn, may prompt early intervention and preservation of the allograft. Three tubes of blood will be drawn twice, 8-12 weeks apart, during clinic or standard of care dialysis visits following optimization. Subjects undergoing desensitization will have three tubes of blood drawn seven times over the course of two years for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be listed for solid organ transplant at NU/NMH
* Subjects should be > or = to 18 years of age, either gender
* Subjects should have history of prior sensitization of HLA antigens
* Subjects should have documented antibody specificity previously tested at the transplant immunology lab at NU
* Subjects should be capable of understanding the study, consents, HIPAA process and be able to give informed consent.

Exclusion Criteria:

* Subjects younger than 18 years of age
* Subjects with no sensitization history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any kidney, pancreas or heart transplant waitlisted subjects > or = to 18 years of age, and of either gender. Subjects must be capable of understanding the study, informed consent form, HIPPA process, and be willing to give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To optimize an in-vitro assay to enumerate HLA-specific memory B cells in order to monitor efficacy of desensitization protocols. | Enrollment (baseline), midpoint of desensitization (only if receiving high dose IVIg); prior to transplant; 3, 6, 12 and 24 months post-transplant.
  B cells will be tested for their ability to produce IgG and tetanus antibodies (as controls) and HLA specific antibodies corresponding to those detected by the flow PRA assay. In subjects not undergoing desensitization, 3 tubes (30 ml) of blood will be drawn twice (total of 60 ml blood taken) 8-12 weeks apart. In subjects undergoing desensitization 3 tubes (30 ml) of blood will be taken at 7 points; enrollment, anticipated midpoint of desensitization, prior to transplant, 3, 6, 12 and 24 Months post-transplant (total of 210 ml blood taken).

SECONDARY OUTCOMES:
Evaluate the relationships between antibody strength, measured by flow cytometry, number of memory B cells in circulation of highly sensitized patients awaiting organ transplant or undergoing desensitization procedures to facilitate organ transplant. | Enrollment (baseline), midpoint of desensitization (only if receiving high dose IVIg); prior to transplant; 3, 6, 12 and 24 months post-transplant.
  B cells will be tested unstimulalated or stimulated with a cocktail of CpG, anti-CD40-L, IL-10 and IL-4.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Tambur, DMD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States